CLINICAL TRIAL: NCT05019651
Title: Acceptability and Feasibility of Apollo Wearable System, Tuned Vibroacoustic Stimulation (TVS) in Veterans With a History of Post-traumatic Stress Disorder (PTSD)
Brief Title: Acceptability and Feasibility of Apollo in Veterans With a History of PTSD
Acronym: Apollo PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisa Brenner (U.S. Federal Agency)
Collaborators: Apollo Neuroscience (Unknown)
Responsible Party: Sponsor-Investigator, Lisa Brenner, Director, Rocky Mountain Mental Illness Research, Education, and Clinical Center, VA Eastern Colorado Health Care System
Organization: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-2268
Record Dates: First submitted 2021-07-16; First posted 2021-08-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: PTSD
Keywords: Stress; Heart Rate Variability; Microbiome
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Apollo Wearable System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm- Apollo Wearable System (Experimental): Apollo Device TVS (10-200 Hz) attached to the subject's wrist or ankle via a commercially available wearable vibration technology can deliver TVS (Transcutaneous Vibratory Stimulation). The intensity will be targeted for the sensory threshold (the level at which the vibration is just noticeable) as this is where the TVS seems to be most effective from prior studies. Similar vibratory stimuli have been demonstrated to be safe in the literature.10-14 The intensity of the vibration will be adjusted to the subjects' comfort and can be controlled by the subject at any time.
  Interventions: Device: Apollo Wearable System

INTERVENTIONS:
Device: Apollo Wearable System — Participants will be provided with the Apollo wearable device and asked to install the study mobile application on their mobile phone. Participants will use the Apollo for at least 30 minutes after waking up in the morning and at least 30 minutes before bed on the corresponding settings for those times of day. They will be given the Apollo Device TVS (10-200 Hz) to borrow which they will be instructed to wear for 6 +/- 2 weeks. They will be asked to continue to wear the device until all study data is collected.

SUMMARY:
The proposed investigation is an open label pilot study intended to establish the acceptability and feasibility of the Apollo in a population of Veterans. Exploratory data regarding biological signatures will also be collected.

DETAILED DESCRIPTION:
Evaluation of Apollo requires a stepwise process in which initial aims are geared towards identifying biological signatures versus diagnosing, treating, mitigating or curing any conditions. Towards the end of identifying potential biological signatures, we hypothesize the following. 1) Participants who use the Apollo will have an attenuated physiological stress response as measured by improved heart rate variability (HRV) compared to baseline. 2) Participants who use Apollo will have attenuated perceived psychological stress measured by lower scores on psychological correlates of acute stress when compared to baseline

ELIGIBILITY:
Inclusion Criteria:

1. Veterans eligible to receive care by a VA provider
2. History of at least one deployment in support of Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND)
3. Current diagnosis of PTSD per the Clinician Administered PTSD Scale-5 (CAPS-5)
4. Willingness to wear the Apollo daily and to comply with study protocol
5. Android or Apple smart phone on which the participant can download the Apollo mobile app
6. Age between 18 and 65
7. Ability to provide informed consent

Exclusion Criteria:

1. Inability to adequately respond to questions regarding the informed consent procedure
2. Currently involved in the criminal justice system as a prisoner or ward of the state
3. Current (past month) alcohol or substance abuse or dependence
4. Lifetime history of bipolar disorder, psychosis, or delusional disorders
5. Lifetime history of oppositional defiant disorder or anti-social personality disorder
6. Pregnancy
7. Recent medication changes in the past 4 weeks
8. A current beta blocker prescription (other than prazosin)
9. Active untreated visual impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability via Credibility Scale | 6 +/- 2 weeks
  The Credibility Scale is a three-item questionnaire that will be used to assess patients' sense of the Apollo Wearable Device credibility.
Acceptability via Expectancy Scale | 6 +/- 2 weeks
  The Credibility Scale is a two-item questionnaire that will be used to assess patients' expectations of the Apollo Wearable Device.
Acceptability via Client Satisfaction Questionnaire (CSQ) | 6 +/- 2 weeks
  Client Satisfaction Questionnaire (CSQ) is an eight-item questionnaire that will be used to assess patients' satisfaction with the intervention. The CSQ has good reliability and validity and has frequently been used to evaluate community mental health care.
Acceptability via Narrative Evaluation of Intervention Interview (NEII) | 6 +/- 2 weeks
  Narrative Evaluation of Intervention Interview (NEII) is a 16-item semi-structured interview that is designed to help participants evaluate and describe the process and outcome of an intervention.
Feasibility via Credibility Scale | 6 +/- 2 weeks
  The Credibility Scale is a three-item questionnaire that will be used to assess patients' sense of the Apollo Wearable Device credibility.
Feasibility via via Expectancy Scale | 6 +/- 2 weeks
  The Credibility Scale is a two-item questionnaire that will be used to assess patients' expectations of the Apollo Wearable Device.
Feasibility via Client Satisfaction Questionnaire (CSQ) | 6 +/- 2 weeks
  Client Satisfaction Questionnaire (CSQ) is an eight-item questionnaire that will be used to assess patients' satisfaction with the intervention. The CSQ has good reliability and validity and has frequently been used to evaluate community mental health care.
Feasibility via Narrative Evaluation of Intervention Interview (NEII) | 6 +/- 2 weeks
  Feasibility will be aNarrative Evaluation of Intervention Interview (NEII) is a 16-item semi-structured interview that is designed to help participants evaluate and describe the process and outcome of an intervention. ssessed using the Credibility/Expectancy Scales, Client Satisfaction Questionnaire (CSQ), and the Narrative Evaluation of Intervention Interview (NEII).

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Colorado Health Care System (ECHCS), Aurora, Colorado, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT05019651/ICF_001.pdf